CLINICAL TRIAL: NCT05269602
Title: The Diagnostic Role of Adding the Hoffman Reflex Study for L5 Radiculopathy in the Electrodiagnostic Laboratory
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hasan Kara, Assistant professor, physiatrist, TC Erciyes University
Other Study IDs: HKara1
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Radiculopathy; Hoffman's Reflex
Keywords: Electrodiagnosis
MeSH Terms: conditions — Radiculopathy; Reflex, Abnormal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- L5 Radiculopathy: Patients who have Lumbar 5 root compression with the Magnetic Resonance İmaging
- S1 Radiculopathy: Patients who have Sacral 1 root compression with the Magnetic Resonance İmaging

SUMMARY:
The H-reflex is one of the most popular topics in reflexology and one of the late responses involved in routine nerve conduction studies in the electromyography (EMG) laboratory. The H-reflex is generally recorded from the gastrocnemius-soleus muscles (tibial H-reflex) by stimulating the tibial nerve in the lower extremity. Tibial H-reflex is a sensitive measurement for examining S1 radiculopathy. Although there are plenty of studies related to the Soleus muscle registered H-reflex in S1 radiculopathy in the literature, there is no study in which the H-reflex is used in L5 muscles in diagnosing L5 radiculopathies. The aim of this study is to investigate the effectiveness of the H-reflex by using a different method in the distinction between L5 and S1 radiculopathies.

DETAILED DESCRIPTION:
The H-reflex is one of the most popular topics in reflexology and one of the late responses involved in routine nerve conduction studies in the electromyography (EMG) laboratory. The H-reflex is generally recorded from the gastrocnemius-soleus muscles (tibial H-reflex) by stimulating the tibial nerve in the lower extremity. Tibial H-reflex is a sensitive measurement for examining S1 radiculopathy.

Hoffman et al. developed a method for simultaneously evaluating the H-reflex obtained from different muscles with single peripheral nerve stimulation. With this method, H-reflex measurement can be done in three leg muscles, including the tibialis anterior, peroneus longus, and soleus with sciatic nerve stimulation. Thus, the L5 and S1 roots can be evaluated separately with a single stimulation.

Although there are plenty of studies related to the Soleus muscle registered H-reflex in S1 radiculopathy in the literature, there is no study in which the H-reflex is used in L5 muscles in diagnosing L5 radiculopathies. The aim of this study is to investigate the effectiveness of the H-reflex by using a different method in the distinction between L5 and S1 radiculopathies.

The H-reflex was evaluated simultaneously using the method developed by Hoffman et al. using superficial recording electrodes in a 3-channel way from the Tibialis anterior, Peroneus Longus, and Soleus muscles.

Latency was recorded when the maximum H-reflex amplitude was obtained. The onset H-reflex latency was marked and measured for each muscle. The patients were evaluated according to EMG and magnetic resonance imaging findings. The latency of the H-reflex was compared with the contralateral extremity in each group.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* Low back pain for at least three months
* Radicular pain in one extremity, disc herniation that matches painful dermatome and root compression in MRI(L5 or S1 root compression)
* MRI and physical examination findings compatible with root compression
* No contraindications to EMG.

Exclusion Criteria:

* Bilateral radicular symptoms
* Multiple levels of radiculopathy
* Diabetes
* Polyneuropathy
* Rheumatic diseases
* History of malignancies
* Lumbosacral region spine surgery
* Lumbar spinal stenosis
* Spondylolisthesis
* Previous peripheral neuropathy in the lower extremities
* Different causes of radiculopathy other than disc herniation (e.g. tumor, osteophyte, facet hypertrophy and other)
* Central system disorders
* Muscular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 58 patients admitted applied to the outpatient clinics due to unilateral radicular back pain and who had L5 or S1 root compression in magnetic resonance imaging (MRI) participated in this study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The Hoffman reflex latency | 1 day
  The Hoffman reflex latency evaluated after electromyography

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University Faculty of Medicine, Ankara, Besevler
  - Selcuk University Faculty of Medicine, Konya, Selcuklu

IPD SHARING:
Plan to Share IPD: Undecided